CLINICAL TRIAL: NCT02091063
Title: A Study of the Selective HDAC6 Inhibitor, ACY-1215, for the Treatment of Patients With Relapsed or Refractory Lymphoid Malignancies
Brief Title: ACY-1215 for Relapsed/Refractory Lymphoid Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Jennifer Amengual (Other)
Collaborators: Acetylon Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Amengual, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAM4054
Record Dates: First submitted 2014-03-14; First posted 2014-03-19 (Estimated); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Lymphoma; Lymphoid Malignancies
Keywords: hematologic malignancies; hodgkin; hodgkins; non-hodgkin; non-hodgkins; mantle cell lymphoma; follicular; lymphoma; lymphoid malignancies
MeSH Terms: conditions — Lymphoma; Hematologic Neoplasms; Lymphoma, Mantle-Cell | interventions — ricolinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase Ib and II: ACY-1215 (Experimental): Participants will receive Phase Ib Arm A: ACY-1215 QD or Arm B: ACY-1215 BID. Once Phase I dosing schedule has been determined. 160 mg BID dosing will be administered for Phase II.
  Interventions: Drug: ACY-1215

INTERVENTIONS:
Drug: ACY-1215 — All patients will take the oral ACY-1215 160mg for 28 consecutive days on a 28-day treatment cycle. Each dose will be administered at least 1 hour after ingestion of food and followed by at least 4 ounces of water. Patients will be instructed not to ingest food or other oral medication for at least 2 hours after each ACY-1215 dose.
  Other Names: Ricolinostat

SUMMARY:
This will be an open-label, single agent, multi-institutional phase Ib/II study of ACY-1215 for the treatment of patients with relapsed or refractory lymphoid malignancies. The target population will include patients with histologically confirmed relapsed or refractory non-Hodgkin's lymphoma or Hodgkin's lymphoma, with an expansion cohort of patients with mantle cell lymphoma.

The phase Ib will be conducted to determine the safety and tolerability of two dosing schedules of ACY-1215 monotherapy in patients with lymphoid malignancies. Patients will be accrued simultaneously to two dose cohorts (Arm A and Arm B) of ACY-1215. Selection into each cohort will occur by alternation. All patients will take the prescribed dose of ACY-1215 orally for 28 consecutive days. Patients enrolled into Arm A will take ACY-1215 160 mg daily (QD), whereas patients enrolled into Arm B will take ACY-1215 160 mg twice daily (BID). ACY-1215 will be supplied as a liquid for oral administration (PO). Each dose will be administered at least 1 hour after ingestion of food followed by at least 4 ounces of water. Patients will be instructed not to ingest food or other oral medication for at least 2 hours after each ACY-1215 dose. Frequency in phase II will be determined based on Phase Ib results.

DETAILED DESCRIPTION:
The emergence of epigenetic therapies has identified pan-class deacetylase (DAC) inhibitors as effective therapeutic agents for the treatment of lymphoma. While pan-class DAC inhibitors have led to FDA indications, clinical activity has been limited to the T-cell derived malignancies. The mechanism of action remains largely unknown and off-target effects lead to side effects including fatigue, gastrointestinal disturbances, and cytopenias. Recently, the development of isoform selective DAC inhibitors have opened the opportunity to investigate their mechanism. It is now recognized that DAC inhibitors not only have epigenetic properties, but have direct effects on transcription factors (p53), oncogenes (Bcl6), and protein degradation pathways (aggresome). Proteolysis occurs primarily through the ubiquitin-proteosome pathway. In states where this pathway is physiologically overwhelmed or therapeutically inhibited, the aggresome sequesters proteins for degradation. DAC6 is a class IIb deacetylase that facilitates misfolded protein transport to the aggresome for proteosome-independent proteolysis. Inhibition of the aggresome activates the unfolded protein response (UPR) pathway, a cellular quality control mechanism with two primary functions: (1) to promote survival during cellular endoplasmic reticulum (ER) stress by chaperoning proteins back for re-folding and halting further transcription until homeostasis is restored and (2) to signal CCAAT/enhancer binding protein (C/EBP)-homologous protein (CHOP) mediated apoptosis when homeostasis cannot be reestablished[9]. While most cells depend on both branches of the UPR to coordinate protein folding, lymphocytes physiologically down-regulate the UPR-apoptosis pathway, specifically CHOP, to allow for generation of high affinity antibodies. In addition to initiating genetic abnormalities (translocations and point mutations) lymphomas inherit this biology, and thus gain a survival advantage.

It has been shown ACY-1215, an Histone Deacetylase 6 (HDAC6)-selective, orally active small-molecule enzyme inhibitor has had single agent activity in a panel of lymphoma cell lines and mouse models, and marked synergistic activity with several agents such as bortezomib, carfilzomib, and ibrutinib, unpublished data. ACY-1215 has been studied in vivo in models of multiple myeloma and lymphoma with marked activity both as a single agent and in combination with bortezomib. Therefore ACY-1215 will be investigated for treatment of lymphoma as a single agent leading to future studies evaluating its effects in combination with other targeted agents known to be active in lymphoma and synergistic with ACY-1215.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed relapsed or refractory non-Hodgkin's lymphoma or Hodgkin's lymphoma (World Health Organization criteria), for which they are unwilling or unable to undergo an autologous stem cell transplant. Patients may have relapsed after prior stem cell transplant.
* Must have received first line chemotherapy. No upper limit to number of prior therapies.
* Patients must have measurable disease.
* Patients must be age ≥ 18.
* Patient has a Karnofsky Performance Status score of ≥70 or Eastern Cooperative Oncology Group (ECOG) performance status score of ≤2
* The patient or the patient's legal representative is able to understand the risks of the study and provide signed informed consent and authorization to use protected health information (in accordance with national and local privacy regulations).
* Patient has adequate bone marrow reserve, as evidenced by:

  * Absolute neutrophil count (ANC) of ≥1.0x109/L.
  * Platelet count of ≥50x109/L.
* Patient has adequate renal function, as evidenced by a creatinine within the institutional limits of normal or a calculated creatinine clearance of ≥30 mL/min according to the Cockcroft-Gault equation.
* Patient has adequate hepatic function, as evidenced by serum bilirubin values <2.0 mg/dL and serum alanine transaminase (ALT) and/or aspartate transaminase (AST) values <3 × the upper limit of normal (ULN) of the local laboratory reference range. (Patients with isolated elevations in alkaline phosphatase (ALP) <5 × ULN in the presence of bony disease are not excluded from participating in the study.)
* Females of childbearing potential must have a negative urine or serum pregnancy test within 7 days of (C1D1) and have adequate contraception. (A female is considered to be not of childbearing potential if she has undergone bilateral oophorectomy or if she has been menopausal without a menstrual period for 12 consecutive months.)

Exclusion Criteria:

* Prior Therapy

  1. Patients who have had chemotherapy or radiotherapy within 2 weeks of study drug treatment or those who have not recovered from adverse events due to agents administered
  2. Systemic steroids that have not been stabilized to the equivalent of ≤10 mg/day prednisone during the 7 days prior to the start of the study drugs.
  3. No monoclonal antibody within 3 months unless evidence of disease progression.
* Patients may not be receiving any other investigational agents.
* Patients with known central nervous system metastases, including lymphomatous meningitis
* Any known cardiac abnormalities such as:

  * Congenital long QT syndrome
  * Corrected QT (QTc) interval ≥ 500 milliseconds;
* Uncontrolled inter-current illness
* Pregnant or nursing women
* Patient is known to be Human Immunodeficiency Virus (HIV)-positive
* Active Hepatitis A, Hepatitis B, or Hepatitis C infection
* Patient has a history of surgery that would interfere with the administration or absorption of the oral study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Amengual, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Moffit Cancer Center, Tampa, Florida
  - Columbia University Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- ACY-1215: 160 mg Once Daily (Phase 1): Cohort 1: Participants were administered ACY-1215 orally once a day for 28 days total.
- ACY-1215: 160 mg Twice Daily (Phase 1): Cohort 2: Participants were administered ACY-1215 orally twice a day for 28 days total.
- ACY-1215: 160 mg Twice Daily (Expansion) (Phase 1): Safety Expansion Cohort: Participants were administered ACY-1215 orally twice a day for 28 days total.
- ACY-1215: 160 mg Twice Daily (Phase 2): Participants were administered ACY-1215 orally twice a day for 28 days total.
Period: Cohort 1: 160 mg Once Daily (Phase 1)
Arm/Group | ACY-1215: 160 mg Once Daily (Phase 1) | ACY-1215: 160 mg Twice Daily (Phase 1) | ACY-1215: 160 mg Twice Daily (Expansion) (Phase 1) | ACY-1215: 160 mg Twice Daily (Phase 2)
Started | 3 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Cohort 2: 160 mg Twice Daily (Phase 1)
Arm/Group | ACY-1215: 160 mg Once Daily (Phase 1) | ACY-1215: 160 mg Twice Daily (Phase 1) | ACY-1215: 160 mg Twice Daily (Expansion) (Phase 1) | ACY-1215: 160 mg Twice Daily (Phase 2)
Started | 0 | 6 | 0 | 0
Completed | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Expansion: 160 mg Twice Daily (Phase 1)
Arm/Group | ACY-1215: 160 mg Once Daily (Phase 1) | ACY-1215: 160 mg Twice Daily (Phase 1) | ACY-1215: 160 mg Twice Daily (Expansion) (Phase 1) | ACY-1215: 160 mg Twice Daily (Phase 2)
Started | 0 | 0 | 4 | 0
Completed | 0 | 0 | 4 | 0
Not Completed | 0 | 0 | 0 | 0
Period: 160 mg Twice Daily (Phase 2)
Arm/Group | ACY-1215: 160 mg Once Daily (Phase 1) | ACY-1215: 160 mg Twice Daily (Phase 1) | ACY-1215: 160 mg Twice Daily (Expansion) (Phase 1) | ACY-1215: 160 mg Twice Daily (Phase 2)
Started | 0 | 0 | 0 | 8
Completed | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All baseline characteristics were collected from the study participants agnostic to their Arm assignment. Baseline characteristics were NOT collected per dose level thus cannot be reported per dose level.
Groups:
- All Participants: Includes participants treated with ACY-1215.
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 55 [24 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16
  Black or African American | 4
  Asian | 1
Disease type [Count of Participants; unit: Participants]
  Hodgkin's Lymphoma | 7
  Diffuse large B-cell Lymphoma (DLBCL) | 5
  T-cell Lymphoma | 4
  Marginal Zone Lymphoma (MZL) | 2
  Mantle Cell Lymphoma (MCL) | 1
  Follicular Lymphoma | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experience a Dose-limiting Toxicity (DLT)
Description: This is designed to establish the safety of 2 dose schedules of ACY-1215 in patients with relapsed or refractory lymphoid malignancies treated with ACY-1215. If more than 1/3 or 2/6 patients experience a DLT in Phase I, there will be no expansion.
Time Frame: Up to 1 year
Population: Data was not collected due to early termination of study, therefore data cannot be analyzed or reported.
Arm/Group | Phase Ib and II: ACY-1215
Number analyzed (Participants) | 0

2. Primary Outcome: Objective Response Rate
Description: The anti-tumor activity of ACY-1215 will be measured by the number of subjects with the response rate in Phase II: complete response [CR] and partial response [PR].
  Complete Response (CR) - Disappearance of all non-target lesions by PET/CT. Nodal Mass: (a) FDG-avid or PET positive prior to therapy; mass of any size permitted if PET negative or (b) Variably FDG-avid or PET negative; regression to normal size on CT. Spleen/Liver: Not palpable, nodules disappeared.
  Partial Response (PR) - Regression of measurable disease and no new sites. Nodal Mass: 50% decrease in SPD of up to 6 largest dominant masses; no increase in size of other nodes, (a) FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site; (b) Variably FDG-avid or PET negative; regression on CT. Spleen/Liver: 50% decrease in SPD of nodules.
Time Frame: Up to 3 years
Population: Data was not collected due to early termination of study, therefore data cannot be analyzed or reported.
Arm/Group | Phase Ib and II: ACY-1215
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: All adverse events were reported/collected from the study participants agnostic to their Arm assignment. Adverse events were NOT collected per dose level thus cannot be reported per dose level.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 1/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 21/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=21)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Confusion (General disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 16 (16)
Fatigue (General disorders) | 9 (9)
Nausea (General disorders) | 13 (13)
Vomiting (General disorders) | 8 (8)
Creatinine increased (Hepatobiliary disorders) | 5 (5)
Hyperkalemia (Blood and lymphatic system disorders) | 4 (4)
Anorexia (General disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fever (General disorders) | 3 (3)
Headache (General disorders) | 3 (3)
Hypercalcemia (Blood and lymphatic system disorders) | 3 (3)
Pain (General disorders) | 9 (9)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 3 (3)
Upper respiratory infection (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT02091063/Prot_SAP_000.pdf